CLINICAL TRIAL: NCT05044273
Title: Evaluation of Effectiveness and Safety of Synergy™ XD Stent and Synergy Megatron™ Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of Synergy XD and Synergy Megatron™ Stent
Acronym: IRIS SynergyXD
Status: Recruiting | Type: Observational
Sponsor: Jung-min Ahn (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Jung-min Ahn, Assistant professor of Medicine, Division of Cardiology, Department of Internal Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2021-02
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Coronary Disease
Keywords: drug eluting stent; percutaneous coronary intervention; real world
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease
  Interventions: Device: Synergy XD stent or Synergy Megatron™ Stent

INTERVENTIONS:
Device: Synergy XD stent or Synergy Megatron™ Stent — Percutaneous coronary intervention with Synergy XD stent or Synergy Megatron™ Stent

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of Synergy XD stent and Synergy Megatron™ Stent in the "real world" daily practice as compared with the other drug-eluting stents.

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, open-label registry to compare the effectiveness and safety of Synergy XD stent and Synergy Megatron™ Stents versus other drug-eluting stents (DES) in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients receiving Synergy XD stent(s) or Synergy Megatron™ stent(s).
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other drug-eluting stents (DESs)
* Terminal illness with life-expectancy ≤1 year.
* Patients with cardiogenic shock

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Synergy XD stent or Synergy Megatron™ stent
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The composite event rate of death, non-fatal myocardial infarction, or target vessel revascularization | 1 year
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
The event rate of all death | 5-year
The event rate of cardiac death | 5-year
The event rate of myocardial infarction | 5-year
The composite event rate of death or myocardial infarction | 5-year
The composite event rate of cardiac death or myocardial infarction | 5-year
The event rate of target-vessel revascularization | 5-year
The event rate of target-lesion revascularization | 5-year
The event rate of stent thrombosis | 5-year
  According to Academic Research Consortium(ARC) criteria
The event rate of stroke | 5-year
The event rate of procedural success | 3 days
  Defined as achievement of final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave myocardial infarction, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (22):
- South Korea (22):
  - Hallym University Medical Center, Anyang
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje university Pusan Paik hospital, Busan
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Samsung Changwon Hospital, Changwon
  - Keimyung University Dongsan Medical Center, Daegu
  - Veterans Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Seoul university Bundang hospital, Seongnam
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided